CLINICAL TRIAL: NCT00326872
Title: A Phase II Study of AZD2171 in Adult Patients With Neurofibromatosis Type 1 and Extensive Plexiform and Paraspinal Neurofibromas
Brief Title: AZD2171 in Treating Patients With Neurofibromatosis Type 1 and Plexiform Neurofibroma and/or Neurofibroma Near the Spine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual prior to interim analysis.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00128; NCI-2009-00128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC047F; CDR0000475761; MC047F (Other: Mayo Clinic); 7133 (Other: CTEP); N01CM17104 (NIH); N01CM62205 (NIH); P30CA015083 (NIH); NCT01646970 (obsolete NCT alias); NCT01664390 (obsolete NCT alias)
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibroma; Spinal Cord Neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Treatment repeats every 28 days for 26 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue treatment beyond 26 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, prior to course 2, prior to course 4, and every 6 courses thereafter.
  Interventions: Drug: Cediranib Maleate

INTERVENTIONS:
Drug: Cediranib Maleate
  Other Names: AZD2171; AZD2171 Maleate; Recentin

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with neurofibromatosis type 1 and plexiform neurofibroma and/or neurofibroma near the spine. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of AZD2171, in terms of volume change in target tumors by 3-dimensional magnetic resonance imaging (3D MRI).

II. Describe and define the toxicities of AZD2171 in these patients.

SECONDARY OBJECTIVES:

I. Assess the value of 3D MRI data analysis in evaluating plexiform or paraspinal neurofibromas compared to conventional 2-dimensional MRI data analysis.

II. Assess the value of delayed contrast-enhanced MRI (DCE-MRI) in determining changes in vascularity of neurofibromas before and during treatment. III. Assess the quality of life of patients treated with AZD2171. IV. Evaluate the effect of AZD2171 on biological changes of human neurofibroma by comparing pre- and post-treatment specimens from patients involved in this trial or, alternatively, by evaluating the effect of AZD2171 on human tumor grafts in experimental animals.

V. Evaluate relevant pharmacodynamic markers (circulating endothelial cells [CECs] and vascular endothelial growth factor-2 [VEGF2] levels) and pharmacogenetics analyses (variation in kdr/flk-1 and other genes) in response to AZD2171.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor location (peripheral vs paraspinal plexiform neurofibroma). Patients receive oral AZD2171 once daily on days 1-28.

Treatment repeats every 28 days for 26 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue treatment beyond 26 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, prior to course 2, prior to course 4, and every 6 courses thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis* of neurofibromatosis type 1 (NF1) and extensive plexiform and/or paraspinal neurofibromasproducing pain (not controlled by use of over-the-counter medications), progressive neurologic deficit, or significant neurologic consequenceswith continuous tumor growth

  * Extensive paraspinal neurofibroma defined as a neurofibroma that involves multiple neural roots at ≥ 3 spinal levels with connection between the levels or extending laterally along the nerves

    * Symptomatic neurofibromas at < 3 spinal levels, but surgical treatment is not possible, allowed
* Meets ≥ 2 diagnostic criteria for NF1, including the following:

  * Six or more café-au-lait spots (≥ 1.5 cm in postpubertal patients)
  * Freckling in the axilla or groin
  * Optic glioma
  * Two or more Lisch nodules
  * Distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia orthinning of long-bone cortex)
  * First-degree relative with NF1
* Patients with documented mutation in neurofibromin gene with onlysymptomatic plexiform and/or paraspinal neurofibroma who do not fulfill the above clinical criteria are eligible
* Measurable disease, defined as ≥ 1 lesion whose longest diameter can beaccurately measured as 8.0 cm^3 with 3-dimensional (3D) MRI

  * Skin lesions are consideredmeasurable (e.g., plexiform neurofibromas), but MRI imaging still required for 3D measurement
* Patients with symptomatic neurofibroma, in whom surgery is not feasible, who refuse surgery or are not goodsurgical candidates due to high risk of damage to vital structures or spinal cordinjury are eligible
* No evidence of progressive optic glioma, malignant glioma, malignant peripheralnerve sheath tumor, or other cancer requiring treatment with chemotherapy orradiotherapy
* ECOG performance status 0-3
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin normal (patients with Gilbert's syndrome allowed despite elevated bilirubin)
* Alkaline phosphatase normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Thyroid-stimulating hormone and free thyroxin normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Ejection fraction ≥ 50% by echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other uncontrolled, serious medical condition that would preclude study participation, including any of the following:

  * Cardiac arrhythmia
  * Diabetes
  * Serious infection
  * Significant cardiac, pulmonary, hepatic, or other organ dysfunction
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergic reactions attributed to compounds of similar chemical orbiologic composition to AZD2171
* No New York Heart Association class III or IV disease

  * Class II disease controlled with treatment and increased monitoring allowed
* No systolic blood pressure (BP) > 130 mm Hg and diastolic BP > 90 mm Hg
* No history of familial long QT syndrome
* Mean QTc ≤ 470 msec (with Bazett's correction) by EKG
* QTc prolongation ≤ 500 msec
* No other significant ECG abnormality within the past 14 days
* See Disease Characteristics
* More than 30 days since prior investigational agents
* More than 4 weeks since prior radiotherapy, chemotherapy, hormonal therapy directed at thetumor, immunotherapy, biologic therapy (e.g., interferon), or majorsurgery
* No concurrent medication that may markedly affect renal function (e.g., vancomycin, amphotericin, or pentamidine)
* No concurrent CYP interactive medications
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent use of drugs or biologics with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-05; Primary Completion 2011-08-21 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dusica Babovic-Vuksanovic, Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Howard University Hospital, Washington D.C., District of Columbia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Case Western Reserve University, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 8/29/2006 until 7/31/2009, 26 patients were accrued.
Pre-assignment Details: All 26 patients accrued were evaluable for the primary endpoint.
Groups:
- Treatment (Cediranib Maleate): Patients receive 30 mg oral AZD2171 once daily on days 1-28. Treatment repeats every 28 days for 26 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease may continue treatment beyond 26 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 34 [19 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Tumor Response (Complete Response [CR] or Partial Response [PR])
Description: Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the volume of target lesions taking as reference the baseline volume.
Time Frame: Baseline to end of treatment, maximum of 26 cycles (28 days/cycle).
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Proportion of patients | 0.0384 [0.002 to 0.216]

2. Secondary Outcome: Survival Time as Measured Using Kaplan-Meier Method
Description: Survival time is defined as the time from registration to death due to any cause.
Time Frame: From registration to death (due to any cause) max 51 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Months | NA [NA to NA] — All 26 patients were alive at last follow-up. Median follow-up time is 24.4 months with a range of 1 to 51 months.

3. Secondary Outcome: Time to Disease Progression as Measured Using Kaplan-Meier Method
Description: Progression (PD): At least a 20% increase in the sum of volumes of target lesions taking as reference the smallest volume recorded since the treatment started or the appearance of one or more new lesions.
  If a patient dies without documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death.
Time Frame: From registration to documentation of disease progression up to 26 cycles (28 days/cycle).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Months | 49.15 [45.76 to NA] — The number of events (n=7) was insufficient to define the upper 95% confidence interval.

4. Secondary Outcome: Duration of Response as Assessed Using the Method of Kaplan-Meier
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed tumor objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented. Duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: From time of confirmed tumor objective response as CR or PR to the date of progression max 51 months
Population: There was only 1 response and due to patient confidentiality we are not reporting this endpoint.
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Treatment Failure as Assessed Using the Method of Kaplan-Meier
Description: Time to treatment failure is defined to be the time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal. If the patient is considered to be a major treatment violation or is taken off study as a non-protocol failure, the patient will be censored on the date they are removed from treatment.
  Time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: From the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal up to 51 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Months | 5.9 [2.6 to 42.3]

6. Secondary Outcome: Reduction in Self Reported Worst Pain Per Cycle.
Description: Reduction in self reported worst pain per cycle as measured by the Worst Pain scale from the North Central Cancer Treatment Group Brief Pain Inventory (short form). The worst pain scale is from 0-10 (10 is worst pain possible). The per-cycle average reduction in worst pain will be analyzed using generalized linear models to account for repeated measures within patients.
Time Frame: At baseline, prior to each subsequent course (q 28+/- 3 days), and at end of treatment up to 51 months
Measure: Mean (Standard Error); unit: units on a scale of 0-10
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
units on a scale of 0-10 | 0.137 (0.0552)

ADVERSE EVENTS:
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 12/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=26)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (7)
Neutrophil count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (4)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=26)
Blood disorder (Blood and lymphatic system disorders) | 6 (51)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (48)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (5)
Palpitations (Cardiac disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 8 (65)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Constipation (Gastrointestinal disorders) | 7 (16)
Diarrhea (Gastrointestinal disorders) | 23 (135)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 12 (37)
Vomiting (Gastrointestinal disorders) | 9 (10)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 16 (125)
Fever (General disorders) | 2 (2)
Flu-like symptoms (General disorders) | 2 (5)
General symptom (General disorders) | 1 (3)
Pain (General disorders) | 3 (4)
Hypersensitivity (Immune system disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Alanine aminotransferase increased (Investigations) | 8 (36)
Alkaline phosphatase increased (Investigations) | 8 (27)
Aspartate aminotransferase increased (Investigations) | 6 (19)
Blood bilirubin increased (Investigations) | 9 (69)
Creatinine increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (10)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 5 (10)
Serum cholesterol increased (Investigations) | 1 (2)
Weight loss (Investigations) | 11 (139)
Anorexia (Metabolism and nutrition disorders) | 6 (13)
Blood glucose increased (Metabolism and nutrition disorders) | 13 (39)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (12)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 3 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (21)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (25)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (18)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (14)
Headache (Nervous system disorders) | 14 (62)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (4)
Peripheral motor neuropathy (Nervous system disorders) | 3 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (44)
Sinus pain (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (11)
Insomnia (Psychiatric disorders) | 5 (20)
Cystitis (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 10 (30)
Irregular menstruation (Reproductive system and breast disorders) | 3 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 6 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (5)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 10 (40)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 11 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less